CLINICAL TRIAL: NCT06786689
Title: Comparing the Efficacy of Weekly Azathioprine Pulse Versus Betamethasone Oral Mini-Pulse in the Treatment of Moderate to Severe Alopecia Areata
Brief Title: To Compare the Efficacy of Weekly Azathioprine Pulse Versus Betamethasone Oral Mini-Pulse in the Treatment of Moderate to Severe Alopecia Areata
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Principal Investigator, Kainat usman, Post Graduate Resident in Dermatology, Sheikh Zayed Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sheikh-ZMC/H
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Alopecia Areata; Alopecia Areata(AA)
Keywords: alopeica areata; azathioprine; oral betamethasone; pulse therapy
MeSH Terms: conditions — Alopecia Areata | interventions — Azathioprine; Betamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Weekly Azathioprine Pulse Therapy (Group A) (Active Comparator): single dose of Tab. Azathioprine 300 mg once weekly
  Interventions: Drug: Azathioprine (AZA)
- Betamethasone Oral Mini Pulse (Group B) (Active Comparator): Tab. Betamethasone 5mg for 2 consecutive days weekly for 3 months
  Interventions: Drug: Betamethasone

INTERVENTIONS:
Drug: Azathioprine (AZA) — weekly single dose of tab azathioprine 300mg
  Arms: Weekly Azathioprine Pulse Therapy (Group A)
Drug: Betamethasone — oral Betamethsone 5mg for 2 consecutive days weekly
  Arms: Betamethasone Oral Mini Pulse (Group B)

SUMMARY:
Alopecia areata (AA) is an autoimmune condition characterized by non-scarring hair loss, ranging from minor patches to complete baldness. Given the variable effectiveness of existing treatments, this study aimed to compare the efficacy of weekly Azathioprine pulse (WAP) therapy against Betamethasone oral mini-pulse (BOMP) therapy in managing moderate to severe AA.

DETAILED DESCRIPTION:
Alopecia areata (AA) is an autoimmune disorder characterized by non-scarring, solitary, or multiple circular or oval patches of hair loss on scalp or other hear bearing areas. These patches often feature "exclamation mark hairs" near their leading edges. It effects all demographics irrespective of age, sex, and ethnicity. Clinically, Alopecia areata can be categorized in various forms depending on extent of involvement, such as patchy hair loss on the scalp, Alopecia Totalis (complete scalp hair loss), or Alopecia Universalis (complete scalp and body hair loss), or less commonly, as band-like hair loss on specific regions of the scalp.

Given the uncertain pathogenesis and course of the disease, the effectiveness of treatment modalities remains unpredictable. Effective treatment must address both the clinical efficacy and safety. Previous studies have reported variable safety profiles, remission, and relapse rates for weekly Azathioprine pulse therapy versus Betamethasone oral mini-pulse therapy, particularly when compared to placebo. However, direct comparisons, especially within our local demographic, are notably lacking. Therefore, this study aimed to bridge the existing gap in literature by offering a comparative evaluation of these therapies in the management of moderate to severe alopecia areata.

ELIGIBILITY:
Inclusion Criteria:

* aged 16-60 years
* scalp area involvement of ≥ 15% by Alopecia Areata

Exclusion Criteria:

* used topical and intralesional treatment within last 1 month,
* received systemic therapy or phototherapy within last three months,
* anemia, leukocytosis, leukopenia, thrombocytopenia, deranged renal and liver function test
* pregnant an lactating females
* patients with contraindications to corticosteroids or Azathioprine

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Severity of Alopecia Tool (SALT) score | Clinical Assessment will be done monthly for 6 months
  photographs of the standard four views of the scalp were captured at initial and follow-up appointments using a 50-megapixel Mobile camera under consistent lighting conditions. The Severity of Alopecia Tool (SALT) score was determined by dividing the scalp into four sections according to their surface areas: the top at 40%, the back at 24%, and each side (left and right) at 18%. The SALT score calculation involved the sum of the percentage of hair loss from the left side (0.18) plus the right side (0.18), the vertex (0.40), and the back (0.24). SALT scores were evaluated at baseline, 12 weeks post-treatment initiation, and 3 months after completion of treatment. Treatment response was determined by using the formula: Percentage of hair regrowth= (SALT score at baseline - SALT score at follow-up) x100 / SALT score at baseline. Treatment response was further divided into 4 categories: Poor response (<25% hair growth improvement from baseline), Moderate response (26-50% improvement), Goo

CONTACTS AND LOCATIONS:
Locations (1):
- Sheikh Zayed Medical College/Hospital, Rahimyarkhan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No